CLINICAL TRIAL: NCT02757950
Title: A Post-marketing, Observational, Retrospective, Cohort Study to Assess the Safety of RefortrixTM (Tdap) When Administered During Pregnancy in a Maternal Immunization Program in Brazil.
Brief Title: A Post-marketing, Observational, Retrospective Study to Assess the Safety of RefortrixTM (Tdap) When Administered During Pregnancy in a Maternal Immunization Program in Brazil.
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 203153
Record Dates: First submitted 2016-04-28; First posted 2016-05-02 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Diphtheria
Keywords: exposed and unexposed cohorts; post-marketing, maternal immunization; neonate related Adverse Events; Congenital anomaly; RefortrixTM; Pregnancy related Adverse Events
MeSH Terms: conditions — Diphtheria; Congenital Abnormalities | interventions — Tetanus Toxoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Exposed cohort: Women, 18-45 years of age at the time of pregnancy, who delivered in the hospital (study centre) from May 2015 and who received one dose of Refortrix during 27 to 36 weeks of pregnancy (or as late as 20 days before delivery due date).
  Interventions: Biological: Combined diphtheria, tetanus and tricomponent acellular pertussis vaccine [Refortrix (Tdap)]
- Unexposed cohort: Women, 18-45 years of age at the time of pregnancy, who delivered in the hospital (study centre) before implementation of the maternal immunization program in Brazil in September 2014 and who did not receive Tdap vaccination during pregnancy.
  Interventions: Biological: Combined diphtheria, tetanus and tricomponent acellular pertussis vaccine [Refortrix (Tdap)]

INTERVENTIONS:
Biological: Combined diphtheria, tetanus and tricomponent acellular pertussis vaccine [Refortrix (Tdap)] — Subjects were included in the Exposed cohort if they received Refortrix as part of the maternal immunization program in Brazil.

SUMMARY:
The purpose of this study is to assess the safety of RefortrixTM (Tdap) when administered during pregnancy in a maternal immunization program in Brazil.

DETAILED DESCRIPTION:
In this retrospective cohort study the safety of RefortrixTM (Tdap) administered during pregnancy as part of the National immunization program in Brazil will be assessed by comparing the risk of pre-defined adverse events before and after introduction of the RefortrixTM (Tdap) maternal immunization program.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 18 and 45 years of age at the time of pregnancy under consideration for the study, who deliver in the study centre.
* Residents of the study area
* Subjects who were compliant with the routine antenatal care including at least one ultrasound assessment report early in the pregnancy.
* Subjects with the complete and relevant medical records available.

Inclusion criteria for the Exposed cohort:

* Subjects who received one dose of Refortrix vaccine in the recommended time period between 27 and 36 completed weeks of pregnancy (or as late as 20 days before delivery due date) as part of the maternal immunization program in Brazil, and according to the program recommendations from May 2015 onwards.
* Subjects with appropriate vaccination records.

Inclusion criteria for the Unexposed cohort:

* Subjects who had delivered in the same hospital (study centre) before 01 September 2014 (September 2012-August 2014) and who did not receive Tdap vaccination during pregnancy to the best knowledge of the investigator.

Exclusion Criteria:

* Subjects who have been transferred to other specialised centres, where their medical records would be inaccessible for the study (private clinics, psychiatric or prison hospitals, other state hospitals, etc).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The subjects who delivered in the study centre from May 2015 onwards will be considered as potentially exposed and those who delivered before September 2014 will be considered as potentially unexposed
Sampling Method: Probability Sample
Enrollment: 2462 (Actual)
Dates: Start 2016-07-14 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Santo André, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sancovski M, Mesaros N, Feng Y, Ceregido MA, Luyts D, De Barros E. Safety of reduced antigen content diphtheria-tetanus-acellular pertussis vaccine when administered during pregnancy as part of the maternal immunization program in Brazil: a single center, observational, retrospective, cohort study. Hum Vaccin Immunother. 2019;15(12):2873-2881. doi: 10.1080/21645515.2019.1627161. Epub 2019 Jun 20. PMID 31216218

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 2462 subjects were enrolled in the study in one center in Brazil.
Period: Overall Study
Arm/Group | Exposed Cohort | Unexposed Cohort
Started | 1203 | 1259
Completed | 1199 | 1248
Not Completed | 4 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exposed Cohort | Unexposed Cohort | Total
Number analyzed (Participants) | 1203 | 1259 | 2462
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.49 (6.15) | 26.28 (6.24) | 26.38 (6.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1203 | 1259 | 2462
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Gestational Diabetes
Description: Gestational diabetes was defined as: Onset or first recognition of abnormal glucose tolerance during pregnancy (the diagnosis is based on administration of glucose challenge test at 24-28 weeks of gestation). Includes Class A1: Euglycaemia achieved with diet and/or exercise and Class A2: Euglycaemia achieved with medication.
Time Frame: After week 27 of pregnancy
Population: Analysis was performed on the Total Cohort (TC), which included all the subjects enrolled in the study with symptom sheets filled-in.
Measure: Count of Participants; unit: Participants
Arm/Group | Exposed Cohort | Unexposed Cohort
Number analyzed (Participants) | 1199 | 1259
Participants | 10 | 22
Statistical Analysis 1: Comparison: Exposed Cohort vs Unexposed Cohort; The analysis contained only the subjects with vaccination date in the Exposed cohort and subjects from the Unexposed cohort; Test type: Other — The comparison of the relative risk with its two sided 95% CI of each primary endpoint between the Exposed cohort and the Unexposed cohort was obtained by means of logistic regression model, using the exposure status as a binary independent variable in the model. Absence of increased relative risk was concluded if the respective 95% CI contained 1; p = 0.1147, Regression, Logistic — A multiple logistic regression model was fitted with a backward selection to identify the possible confounding factors for each of the primary safety event using an alpha level of 0.1; Incidence rate ratio = 0.548, 95% CI 2-sided [0.259 to 1.157]

2. Primary Outcome: Number of Subjects Reporting Pregnancy-related Hypertension, Pre-eclampsia, Eclampsia, and HELLP Syndrome
Description: Pregnancy-related hypertension is defined as:
  Blood pressure systolic higher than (>) 140 and/or diastolic > 90 millimetre of mercury (mmHg), documented in at least two separate measurements after 20 weeks of gestation, without proteinuria or other stigmata of pre-eclampsia, and returning to normal post-partum. Hypertension usually resolves by 12 weeks post-partum, included pre-eclampsia, eclampsia and haemolysis elevated liver enzymes low platelet (HELLP) Syndrome for this study.
Time Frame: After week 27 of pregnancy
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Exposed Cohort | Unexposed Cohort
Number analyzed (Participants) | 1199 | 1259
Participants
  Pregnancy-related hypertension | 11 | 31
  Pre-eclampsia | 10 | 30
  Eclampsia | 2 | 0
  HELLP syndrome | 0 | 1
Statistical Analysis 1: Comparison: Exposed Cohort vs Unexposed Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0155, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Incidence rate ratio = 0.428, 95% CI 2-sided [0.215 to 0.851]

3. Primary Outcome: Number of Subjects Reporting Pregnancy Hemorrhage
Description: Pregnancy vaginal hemorrhage is defined as: excessive blood loss after delivery i.e. estimated blood loss in excess of 500 milliliters (ml) after vaginal delivery and estimated blood loss in excess of 1000 ml after Caesarean delivery. The other symptoms are higher than or equal to (≥) 10 percent (%) drop in hematocrit, need for blood transfusion, symptomatic hypotension, dizziness, pallor and oliguria.
  Vaginal or intrauterine hemorrhage that encompasses antepartum (i.e. bleeding from the genital tract after 24 weeks of gestation), intrapartum, and postpartum bleeding (i.e. within 24 hours post-delivery).
  A major obstetric hemorrhage is defined as blood loss from uterus or genital tract >1500 ml or a decrease.
Time Frame: After week 27 of pregnancy
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Exposed Cohort | Unexposed Cohort
Number analyzed (Participants) | 1199 | 1259
Participants | 4 | 19
Statistical Analysis 1: Comparison: Exposed Cohort vs Unexposed Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0127, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Incidence rate ratio = 0.254, 95% CI 2-sided [0.086 to 0.746]

4. Primary Outcome: Number of Subjects With Pre-specified Neonate-related Outcomes Resulting in Preterm Birth
Description: Preterm birth is defined as: Birth before 37 weeks of gestation.
Time Frame: From week 27 up to week 37 of pregnancy
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Exposed Cohort | Unexposed Cohort
Number analyzed (Participants) | 1199 | 1259
Participants | 64 | 121
Statistical Analysis 1: Comparison: Exposed Cohort vs Unexposed Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0036, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Incidence rate ratio = 0.638, 95% CI 2-sided [0.471 to 0.863]

5. Primary Outcome: Number of Subjects With Pre-specified Neonate-related Outcomes, Resulting in Neonates Small for Their Gestational Age
Description: Small for gestational age is defined as: Birth weight less than (<) 10% for infants of same gestational age and gender in same population.
Time Frame: After week 27 of pregnancy
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Exposed Cohort | Unexposed Cohort
Number analyzed (Participants) | 1199 | 1259
Participants | 69 | 62
Statistical Analysis 1: Comparison: Exposed Cohort vs Unexposed Cohort; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0931, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Incidence rate ratio = 1.342, 95% CI 2-sided [0.952 to 1.890]

6. Secondary Outcome: Number of Subjects Reporting Pregnancy-related Adverse Events (AEs) of Interest/Neonate-related Events up to Delivery
Description: Pregnancy-related AEs of interest and neonate-related events are defined as: premature rupture of membranes, preterm premature rupture of membranes, premature uterine contraction, neonatal death, maternal death, still birth, neonatal hypoxic ischaemic encephalopathy.
Time Frame: After week 27 of pregnancy
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Exposed Cohort | Unexposed Cohort
Number analyzed (Participants) | 1199 | 1259
Participants
  Premature rupture of membranes | 190 | 261
  Preterm premature rupture of membranes | 17 | 36
  Premature uterine contractions | 32 | 54
  Neonatal death | 0 | 8
  Maternal death | 0 | 0
  Still births | 1 | 6
  Neonatal hypoxic ischaemic encephalopathy | 0 | 0

7. Secondary Outcome: Number of Subjects Reporting Cases of Congenital Anomalies in the Neonates
Description: Congenital anomalies include morphological, functional, chromosomal or genetic anomalies, regardless of whether detected at birth or not, the foetus is delivered dead or alive, or defects are identified by prenatal ultrasound, amniocentesis or examination of the products of conception.
Time Frame: From week 27 of pregnancy up to birth
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Exposed Cohort | Unexposed Cohort
Number analyzed (Participants) | 1199 | 1259
Participants | 3 | 22

8. Secondary Outcome: Number of Subjects With Pregnancy-related AEs and Birth Outcomes Per Calendar Year
Description: Pregnancy related AEs include: gestational diabetes, pregnancy-related hypertension, pre-eclampsia, eclampsia, HELLP Syndrome and pregnancy hemorrhage. Birth outcomes include: preterm birth and small for gestational age.
Time Frame: After week 27 of pregnancy
Population: Analysis was performed on the Unexposed Cohort which included women pregnant before implementation of the maternal immunization program, who didn't receive Refortrix, the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Unexposed Cohort
Number analyzed (Participants) | 633
Participants
  Gestational diabetes, Sep2012-Aug2013: number analyzed (Participants) | 615
  Gestational diabetes, Sep2012-Aug2013 | 10
  Gestational diabetes, Sep2013-Aug2014 | 12
  Pregnancy-related hypertension, Sep2012-Aug2013: number analyzed (Participants) | 615
  Pregnancy-related hypertension, Sep2012-Aug2013 | 14
  Pregnancy-related hypertension, Sep2013-Aug2014 | 17
  Vaginal hemorrhage, Sep2012-Aug2013: number analyzed (Participants) | 615
  Vaginal hemorrhage, Sep2012-Aug2013 | 16
  Vaginal hemorrhage, Sep2013-Aug2014 | 3
  Preterm birth, Sep2012-Aug2013: number analyzed (Participants) | 615
  Preterm birth, Sep2012-Aug2013 | 66
  Preterm birth, Sep2013-Aug2014 | 55
  Small for gestational age, Sep2012-Aug2013: number analyzed (Participants) | 615
  Small for gestational age, Sep2012-Aug2013 | 31
  Small for gestational age, Sep2013-Aug2014 | 31
  Pre-Eclampsia, Sep2012-Aug2013: number analyzed (Participants) | 615
  Pre-Eclampsia, Sep2012-Aug2013 | 13
  Pre-Eclampsia, Sep2013-Aug 2014 | 17
  Eclampsia, Sep2012-Aug2013 | 0
  Eclampsia, Sep2013-Aug 2014 | 0
  HELLP Syndrome, Sep2012-Aug2013 | 1
  HELLP Syndrome, Sep2013-Aug 2014 | 0

ADVERSE EVENTS:
Time Frame: Entire study period (From week 27 of pregnancy up to birth).
Description: During this retrospective, observational study safety data was not recorded/collected.
Arm/Group | Unexposed Cohort | Exposed Cohort
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-09-11): https://cdn.clinicaltrials.gov/large-docs/50/NCT02757950/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT02757950/SAP_001.pdf